CLINICAL TRIAL: NCT06122831
Title: A Phase Ib/II Clinical Trial of TQ05105 Tablets Combined With TQB3617 Capsules in the Treatment of Intermediate- and High-risk Myelofibrosis
Brief Title: A Clinical Trial of TQ05105 Tablets Combined With TQB3617 Capsules in the Treatment of Myelofibrosis (MF)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-TQB3617-Ib/II-01
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 Tablets + TQB3617 Capsules (Experimental): TQ05105 Tablets combined with TQB3617 Capsules, orally administered. 21 days as a treatment cycle.
  TQB3617 Capsules, orally administered, 21 days as a treatment cycle.
  Interventions: Drug: TQ05105 Tablets; Drug: TQB3617 Capsules

INTERVENTIONS:
Drug: TQ05105 Tablets — TQ05105 Tablets is a Janus kinase 1 (JAK1) and Janus kinase 2 (JAK2) Inhibitor.
Drug: TQB3617 Capsules — TQB3617 Capsules is a Bromodomain and Extra-Terminal (BET) Inhibitor

SUMMARY:
This is an open, single-arm, multi-center clinical study designed to evaluate the efficacy and safety of TQ05105 Tablets combined with TQB3617 Capsules in patients with intermediate- and high-risk Myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and signed informed consent, good compliance.
* Age: 18 or above (when signing the informed consent form); Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 2; Life expectancy ≥ 24 weeks.
* Patients diagnosed with Primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (post PV MF), or post essential thrombocythemia myelofibrosis (post ET MF)
* According to the dynamic international prognostic scoring system (DIPSS), patients with intermediate or high risk of bone marrow fibrosis were evaluated.
* Within 7 days before the first administration, the symptom score of myeloproliferative neoplasms should meet certain requirements.
* Patients with poor efficacy of JAK inhibitors (for phase Ib and phase II cohort 2, cohort 3)
* Patients who had not received JAK inhibitor treatment (for phase II cohort 1).
* Spleen enlargement.
* Peripheral blood primary cells and bone marrow primary cells were ≤10%.
* No growth factor, colony stimulating factor, thrombopoietin or platelet transfusion was received within 2 weeks before the examination, and the blood routine indexes met the requirements within 7 days before the first administration.
* The Main organ function is normal.
* Men and women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study. Serum human chorionic gonadotrophin (HCG) test is not negative within 7 days before the first administration and must be non-lactating patients.

Exclusion Criteria:

* Patients who have previously received allogeneic stem cell transplantation, or received autologous stem cell transplantation within 3 months before the first administration, or recently planned stem cell transplantation;
* Previous treatment with BET inhibitors combined with JAK inhibitor;
* Patients who have previously undergone splenectomy, or received splenic radiotherapy within 6 months before the first administration;
* Use of any MF medications, any immunomodulators, any immunosuppressive agents, within 2 weeks prior to first administration (There are separate withdrawal requirements for hydroxyurea, JAK inhibitors, androgen drugs, erythropoietin, long-acting recombinant interferon-α, etc.);
* Other malignancies within 3 years prior to first administration or currently present.
* Patients with multiple factors (such as inability to swallow, postoperative gastrointestinal resection, acute and chronic diarrhea, intestinal obstruction, etc.) affecting oral or absorption of drugs;
* Major surgical treatment or significant traumatic injury within 4 weeks prior to first administration;
* Presence of congenital bleeding disorder and congenital coagulopathy;
* Patients who had arterial/venous thrombosis events within 6 months before the first administration.
* Have a history of mental drug abuse, or have a mental disorder.
* Active or uncontrolled severe infection;
* Active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection and HCV RNA positive, or active Corona Virus Disease 2019 (COVID-19) infection;
* Patients with grade III or above congestive heart failure, unstable angina pectoris or myocardial infarction, or arrhythmia requiring treatment, or QT interval prolongation within 6 months before the first administration;
* Unsatisfactory blood pressure control despite standard therapy;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Patients newly diagnosed with pulmonary interstitial fibrosis or drug-related interstitial lung disease within 3 months before the first administration;
* Patients with a history of immunodeficiency disease or organ transplantation;
* Patients with epilepsy requiring treatment;
* Patients who have received Chinese patent medicines with anti-tumor indications specified in the approved drug package insert of China National Medical Products Administration (NMPA) within 2 weeks before the first administration;
* Patients with uncontrolled pleural effusion, pericardial effusion or ascites;
* There was a history of attenuated live vaccine inoculation within 4 weeks before the first administration, or attenuated live vaccine inoculation was planned during the study period.
* People with known hypersensitivity to the study drug and excipients;
* Patients diagnosed as active autoimmune diseases within 2 years before the first administration;
* Those who participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first administration (except JAK inhibitor-related clinical trials).
* According to the judgment of the investigators, some situations seriously endanger the safety of the subjects or affect the subjects to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerance dose (MTD) | Up to 2 years.
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.
Recommended phase II dose (RP2D) | Up to 2 years
  The RP2D is defined as the lower dose level to MTD based on the safety profile.
≥35% reduction in spleen volume (SVR35) | Up to 24 weeks
  The proportion of subjects with a ≥35% reduction in spleen volume from baseline at the end of treatment at week 24.

SECONDARY OUTCOMES:
SVR35 | Up to 120 weeks
  The proportion of subjects with a ≥35% reduction in spleen volume compared to baseline after treatment.
Optimum effective rate | Up to 120 weeks
  The proportion of subjects with at least once spleen volume reduction ≥ 35% from baseline.
Onset time of splenic response | Up to 120 weeks
  The time interval from the first administration to the date when the spleen volume was reduced by ≥ 35 % from baseline.
Duration of maintenance of at least 35% Reduction in Spleen Volume (DoMSR) | Up to 120 weeks
  The time between the date when the spleen volume reduction ≥ 35% from baseline occurs for the first time and the date when the spleen volume reduction is < 35% from baseline.
Myeloproliferative neoplasm - Symptom Assessment Form - Total Symptom Score (MPN-SAF TSS) | Up to 60 weeks
  The proportion of subjects whose total symptom score of MPN-SAF TSS decreased by more than 50% from baseline. MPN-SAF-TSS is an effective tool for evaluating the disease burden of patients with myeloproliferative neoplasms. Each symptom is scored according to the severity, from asymptomatic (0 points) to the most serious (10 points), a total of 10 levels, the sum of 10 symptom scores is MPN-SAF-TSS score. The higher the score, the more severe the symptoms are.
MPN-SAF TSS change | Up to 120 weeks
  The total score of MPN-SAF TSS decreased compared with baseline. MPN-SAF-TSS is an effective tool for evaluating the disease burden of patients with myeloproliferative neoplasms. Each symptom is scored according to the severity, from asymptomatic (0 points) to the most serious (10 points), a total of 10 levels, the sum of 10 symptom scores is MPN-SAF-TSS score. The higher the score, the more severe the symptoms are.
Variant allele frequency (VAF) | Up to 48 weeks
  The proportion of subjects whose VAF decreased compared with baseline.
The proportion of subjects with gene mutation achieving SVR35 | Up to 48 weeks
  The proportion of subjects with gene mutation achieving SVR35
The proportion of subjects with gene mutation whose MPN-SAF TSS scale decreased by ≥ 50% | Up to 48 weeks.
  The proportion of subjects with gene mutation whose MPN-SAF TSS scale decreased by ≥ 50% compared with baseline.
Progression-free survival (PFS) | Up to 120 weeks
  The time interval from the first dose to the date of the occurrence of any of the following events, whichever occurs first:(1) Spleen volume increased by ≥25% compared with the screening period ; (2) Death caused by any cause.
Leukemia free survival (LFS) | Up to 120 weeks
  The time interval from the date of the first dose to the date of any of the following events, whichever occurs first: (1) the date of the first bone marrow smear showing the original cell ≥20% ;(2) The first peripheral blood smear showed that the original cells ≥ 20% and the absolute value of the original cells ≥1×10^9/L and lasted for at least 2 weeks; (3) Death caused by any reason.
Overall Survival (OS) | Up to 120 weeks
  OS is defined as the time from the first time the subject received treatment to death due to any cause.
Incidence of adverse events (AEs) | Baseline up to 120 weeks
  Incidence rate of all adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
Severity of adverse events (AEs) | Baseline up to 120 weeks
  Severity of all adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Cangzhou People's Hosipital, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - North China of Science and Technology University Affiliated Hospital, Tangshan, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Hospital of Harbin, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Tongji College Huazhong Unizersity of Science And Technology, Wuhan, Hubei
  - Wuhan University Zhongnan Hospital, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Public Hospital of Wuxi, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Xi 'An Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi
  - Tai'an City Central Hospital, Tai’an, Shandong
  - Central Hospital Of Minhang District, Shanghai, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - People's Hospital of Tianjin City, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang